CLINICAL TRIAL: NCT00822900
Title: Phase 3 Clinical Trial to Determine if Progesterone Along With Standard Medical Care for Brain Injury is More Effective at Limiting the Amount of Damage Cause by a Traumatic Brain Injury Than Standard Medical Care Alone.
Brief Title: Progesterone for the Treatment of Traumatic Brain Injury III
Acronym: ProTECT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: futility: low conditional power to demonstrate benefit of progesterone
Sponsor: David Wright (Other)
Collaborators: Medical University of South Carolina (Other); Neurological Emergencies Treatment Trials Network (NETT) (Network)
Responsible Party: Sponsor-Investigator, David Wright, Principal Investigator, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00014409; 1RO1 NS062778-01
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Results first posted 2015-07-03 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Traumatic Brain Injury
Keywords: Trauma; Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries; Brain Injuries | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progesterone (Experimental): Following a one hour loading dose of 0.714 mg/kg per infusion pump through a dedicated IV line, the study drug (progesterone) will be administered as a continuous intravenous infusion at 0.5 mg/kg/hr for 71 hours, then tapered over an additional 24 hours. To simplify the infusion protocol, a weight based dosing table will be used by the on-sight pharmacy to mix the correct dose for a 10 cc/hour continuous infusion over the 72 hour steady state period followed by three additional 8-hour decrements (7.5 cc/hr-5.0 cc/hr-2.5 cc/hr) to zero, for a total treatment duration of 96 hour. The progesterone will be combined with a 20% Intralipid mixture for infusion.
  Interventions: Drug: Progesterone
- Placebo (Placebo Comparator): Placebo stock solution was the ethanol diluent required for dissolving progesterone. The volume of placebo to be mixed with intralipid was based on the same mg/kg/hr volume that would be required if PROG had been in the vial. Using an infusion pump through a dedicated IV line - a one hour "loading dose" of placebo plus intralipid was administered as a continuous intravenous infusion for 71 hours, then tapered over an additional 24 hours. To simplify the infusion protocol, a weight based dosing table was used by the on-sight pharmacy to mix the correct "dose" for a 10 cc/hour continuous infusion over the 72 hour steady state period followed by three additional 8-hour decrements (7.5 cc/hr-5.0 cc/hr-2.5 cc/hr) to zero, for a total treatment duration of 96 hour. The placebo will be combined with a 20% Intralipid mixture for infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — Following a one hour loading dose of 0.714 mg/kg per infusion pump through a dedicated IV line, the study drug (progesterone or placebo) will be administered as a continuous intravenous infusion at 0.5 mg/kg/hr for 71 hours, then tapered over an additional 24 hours. To simplify the infusion protocol, a weight based dosing table will be used by the on-sight pharmacy to mix the correct dose for a 10 cc/hour continuous infusion over the 71 hour steady state period followed by three additional 8-hour decrements (7.5 cc/hr-5.0 cc/hr-2.5 cc/hr) to zero, for a total treatment duration of 96 hour. The progesterone/placebo will be combined with a 20% Intralipid mixture for infusion.
  Arms: Progesterone
Drug: Placebo — Placebo stock solution is the ethanol diluent required for dissolving progesterone. The volume of placebo to be mixed with intralipid is based on the mg/kg/hr volume. Using an infusion pump through a dedicated IV line - a one hour "loading dose" of placebo plus intralipid is administered as a continuous intravenous infusion for 71 hours, then tapered over an additional 24 hours.
  Arms: Placebo

SUMMARY:
The ProTECT study will determine if intravenous (IV) progesterone (started within 4 hours of injury and given for a total of 96 hours), is more effective than placebo for treating victims of moderate to severe acute traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe brain injury (GCS 12-4)
* Age 18 years or older
* Blunt, closed head injury
* Study drug initiated within 4 hours of injury

Exclusion Criteria:

* Non-Survivable injury
* Bilateral dilated unresponsive pupils
* Severe intoxication (ETOH > 250 mg %)
* Spinal cord injury with neurological deficits
* Inability to perform activities of daily living prior to injury
* Cardiopulmonary arrest
* Status epilepticus on arrival
* Systolic blood pressure (SBP) < 90 on arrival or for at least 5 minutes prior to enrollment
* O2 Sat < 90 on arrival or for at least 5 minutes prior to enrollment
* Prisoner or ward of state
* Pregnant
* Active breast or reproductive organ cancers
* Known allergy to progesterone or intralipid components (egg yolk)
* Known history of clotting disorder
* Active thromboembolic event
* Concern for inability to follow up at 6 months
* Anyone listed in the Opt out registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 2010-03; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Wright, MD, Principal Investigator — Emory University
Locations (36):
- United States (36):
  - Maricopa Integrated Health System, Phoenix, Arizona
  - Banner Good Samaritan, Phoenix, Arizona
  - Scottsdale Healthcare, Scottsdale, Arizona
  - University of Arizona Medical Center, Tuscon, Arizona
  - Santa Clara Valley Hospital, Palo Alto, California
  - Stanford Medical Center, Palo Alto, California
  - San Francisco General Hospital, San Francisco, California
  - Regional Medical Center-San Jose, San Jose, California
  - Grady Memorial Hospital, Atlanta, Georgia
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Maryland Shock Trauma, Baltimore, Maryland
  - Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Sinai Grace Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Beaumont Royal Oak Hospital, Royal Oak, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Hospital, Robbinsdale, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - St. Johns Mercy Medical Center, St Louis, Missouri
  - Columbia New York Presbyterian Hospital, New York, New York
  - University Hospital, Cincinnatti, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson UniversityHospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Regional Medical Center/Elvis Presley Memorial Trauma Center (The MED), Memphis, Tennessee
  - Austin/Brackenridge, Austin, Texas
  - Memorial Hermann, Houston, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - Virginia Commonwealth, Richmond, Virginia
  - Froedtert East Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Zhao W, Pauls K. Architecture design of a generic centralized adjudication module integrated in a web-based clinical trial management system. Clin Trials. 2016 Apr;13(2):223-33. doi: 10.1177/1740774515611889. Epub 2015 Oct 13. PMID 26464429
- [Derived] Wright DW, Yeatts SD, Silbergleit R, Palesch YY, Hertzberg VS, Frankel M, Goldstein FC, Caveney AF, Howlett-Smith H, Bengelink EM, Manley GT, Merck LH, Janis LS, Barsan WG; NETT Investigators. Very early administration of progesterone for acute traumatic brain injury. N Engl J Med. 2014 Dec 25;371(26):2457-66. doi: 10.1056/NEJMoa1404304. Epub 2014 Dec 10. PMID 25493974

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 882 patients underwent randomization at 49 trauma centers in the United States between April 5, 2010, and October 30, 2013. 442 patients were randomized to Progesterone Arm and 440 were randomized to Placebo Arm.
Period: Overall Study
Arm/Group | Progesterone | Placebo
Started | 442 | 440
Completed | 334 | 347
Not Completed | 108 | 93
Not completed — Withdrawal by Subject | 14 | 14
Not completed — Lost to Follow-up | 9 | 9
Not completed — Death | 83 | 69
Not completed — Became a ward of the state | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Progesterone | Placebo | Total
Number analyzed (Participants) | 442 | 440 | 882
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (18) | 38 (17) | 39 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 114 | 232
  Male | 324 | 326 | 650
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61 | 64 | 125
  Not Hispanic or Latino | 347 | 343 | 690
  Unknown or Not Reported | 34 | 33 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 7
  Asian | 20 | 22 | 42
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 70 | 64 | 134
  White | 330 | 331 | 661
  More than one race | 3 | 6 | 9
  Unknown or Not Reported | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 442 | 440 | 882
Index GCS score at randomization [Number; unit: participants] — The index Glasgow Coma Scale (GCS) score is the highest reliable GCS score documented before randomization.The GCS is scored between 3 and 15, 3 being the worst, and 15 the best. A score of 13 or higher correlates with a mild brain injury, 9 to 12 is a moderate injury and 8 or less a severe brain injury.
  participants
    Moderate | 129 | 125 | 254
    Moderate to severe | 234 | 238 | 472
    Severe | 79 | 77 | 156

OUTCOME MEASURES:

1. Primary Outcome: Favorable Outcome as Determined by the Glasgow Outcome Scale-Extended (GOSE)
Description: A measure of functional recovery: A GOS-E score of 1 indicates death, 2 indicates a vegetative state, 3 or 4 indicates severe disability, 5 or 6 indicates moderate disability, and 7 or 8 indicates good recovery. Favorable outcome was defined via stratified dichotomy based on the severity of the initial injury. For subjects with a severe injury, a GOS-E of 3 or higher were considered to be a favorable outcome; for subjects with moderate-to-severe injury, a GOS-E of 5 or higher was considered to be a favorable outcome; for subjects with a moderate injury, a GOS-E of 7 or higher was considered to be a favorable outcome.
Time Frame: 6 months post randomization
Population: The primary analysis was conducted according to intention to treat.
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 442 | 440
participants
  Favorable Outcome | 213 | 232
  Unfavorable | 201 | 184
  Missing Data | 28 | 24
Statistical Analysis 1: Comparison: Progesterone vs Placebo; Test of null hypothesis (equal proportions of subjects with favorable outcome in progesterone and placebo arms) versus alternative hypothesis (unequal proportions of subjects with favorable outcome in progesterone and placebo arms). Standard multiple imputation methods are used to account for missing data. The primary outcome measure is based on the stratified dichotomy approach; Test type: Superiority or Other; p = 0.35, Regression, Generalized linear; Adjusting for injury severity, sex, and age. the binomial distribution with the log link is used to estimate treatment effect as relative risk; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.85 to 1.06] — A risk ratio (equivalent to the relative risk) of less than 1.00 indicating fewer favorable outcomes in the progesterone group than in the placebo group

2. Secondary Outcome: Mortality
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 442 | 440
participants
  Subjects with events | 83 | 69
  Subjects without events | 359 | 371
Statistical Analysis 1: Comparison: Progesterone vs Placebo; The Cox proportional hazards model is used to compare these curves after adjustment for age, sex and injury severity; Test type: Superiority or Other; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.86 to 1.63] — A hazard ratio of more than 1.00 indicating higher hazard of death from the progesterone group than in the placebo group

3. Secondary Outcome: Disability Rating Scale
Description: A measure of functional impairment, with complete recovery scored a 0 and vegetative state scored a 29.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 442 | 440
units on a scale | 2.9 (4.6) | 3.3 (5.1)

4. Secondary Outcome: Potentially Associated Adverse Events: Phlebitis/Thrombophlebitis
Description: Phlebitis/Thrombophlebitis (not due to infiltration or misplacement of the IV)
Time Frame: within 6 months
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 442 | 440
participants
  Subjects with events | 76 | 25
  Subjects without events | 366 | 415
Statistical Analysis 1: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 3.03, 95% CI 2-sided [1.96 to 4.66] — A risk ratio (equivalent to the relative risk) of more than 1.00 indicating more events in the progesterone group than in the placebo group

5. Secondary Outcome: Potentially Associated Adverse Events: Pulmonary Embolism
Description: Pulmonary embolism - Events were defined based on either positive chest computed tomography (CT) scanning or ventilation/perfusion lung scan (V/Q).
Time Frame: within 6 months
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 442 | 440
participants
  Subjects with events | 10 | 13
  Subjects without events | 432 | 427

6. Secondary Outcome: Potentially Associated Adverse Events: Acute Ischemic Stroke
Description: Acute ischemic stroke - Events were defined based on either positive computed tomography (CT) scanning, magnetic resonance imaging (MRI), or neurologist diagnosis of cerebrovascular accident (CVA)
Time Frame: within 6 months
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 442 | 440
participants
  Subjects with events | 6 | 13
  Subjects without events | 436 | 427

7. Secondary Outcome: Potentially Associated Adverse Events: Deep Venous Thrombosis (DVT)
Description: DVT - Events were defined based on a positive Doppler ultrasound exam
Time Frame: within 6 months
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 442 | 440
participants
  Subjects with events | 50 | 40
  Subjects without events | 392 | 400

8. Secondary Outcome: Potentially Associated Adverse Events: Unexplained Increased Liver-enzyme Level
Description: Unexplained increased liver enzymes (e.g. not due to liver injury ) - Events were defined based on aspartate transaminase (AST) and alanine transaminase (ALT) levels > 500 U/L and/or total bilirubin levels > 2.0 mg/dL.
Time Frame: within 6 months
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 442 | 440
participants
  Subjects with events | 18 | 14
  Subjects without events | 424 | 426

9. Secondary Outcome: Potentially Associated Adverse Events: Sepsis
Description: Sepsis - Events must have met Centers for Disease Control and Prevention (CDC) definition of sepsis. The definition includes that a patient ≤1 year of age has at least 1 of the following clinical signs or symptoms with no other recognized cause: fever (>38°C rectal), hypothermia (<37°C rectal), apnea, or bradycardia, and blood culture not done or no organisms detected in blood and no apparent infection at another site and physician institutes treatment for sepsis.
Time Frame: within 6 months
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 442 | 440
participants
  Subjects with events | 9 | 9
  Subjects without events | 433 | 431

10. Secondary Outcome: Potentially Associated Adverse Events: Pneumonia
Description: Events must have met Centers for Disease Control and Prevention (CDC) definition of pneumonia. There are three specific types of pneumonia: clinically defined pneumonia, pneumonia with specific laboratory findings, and pneumonia in immunocompromised patients. There are specific algorithms to identify each pneumonia, which include x-ray findings, fever with no other cause, leukopenia or leukocytosis, altered mental status with no other cause (adults >70 years old), new onset of purulent sputum, change in character of sputum, increase respiratory secretions, increase suctioning requirements, new onset or worsening cough, dyspnea, tachypnea, rales, bronchial breath sounds, or worsening gas exchange, increased oxygen requirements, or increased ventilator demand). Also, labs can identify pneumonia such as positive growth in blood culture, positive Gram stain, and histopathologic exam evidence.
Time Frame: within 6 months
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 442 | 440
participants
  Subjects with events | 142 | 140
  Subjects without events | 300 | 300

11. Secondary Outcome: Potentially Associated Adverse Events: Central Nervous System (CNS) Infection
Description: CNS infection - Events must have met Centers for Disease Control and Prevention (CDC) definition of CNS infection. The definition includes intracranial infection, Meningitis, ventriculitis, and spinal abscess without meningitis.
Time Frame: within 6 months
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 442 | 440
participants
  Subjects with events | 5 | 3
  Subjects without events | 437 | 437

12. Secondary Outcome: Potentially Associated Adverse Events: Myocardial Infarction (MI)
Description: Myocardial infarction - Events were defined based on serial cardiac enzyme elevation consistent with MI and/or new ST elevation on electrocardiogram (ECG) consistent with MI. Potentially associated adverse events (those events which are included as outcome measures) were specifically defined per the protocol, and the classification of an event as a PAAE was determined by the site. The reported name of the associated event, however, was subject to clinical judgement and case details; these were then further coded by the Principal Investigator. Since these data points do not share the same definition, there is no reason to expect perfect concordance. (For example, the potentially associated adverse event of myocardial infarction may include MedDRA codes other than myocardial infarction.)
Time Frame: within 6 months
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 442 | 440
participants
  Subjects with events | 5 | 5
  Subjects without events | 437 | 435

ADVERSE EVENTS:
Time Frame: Within 6 month after the enrollment.
Description: Preferred terms from the MedDRA vocabulary were assigned by investigators for AE names that did not map to lowest level terms and for those where multiple terms mapped to clinically equivalent events.
Arm/Group | Progesterone | Placebo
Serious Adverse Events (participants affected / at risk) | 246/442 | 251/440
Other Adverse Events (participants affected / at risk) | 332/442 | 330/440
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone (N=442) | Placebo (N=440)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 11 (11) | 7 (7)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 4 (4)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 3 (3) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3) | 3 (3)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (1) | 2 (2)
Device occlusion (General disorders) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Biloma (Hepatobiliary disorders) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 2 (2)
Bacteremia (Infections and infestations) | 7 (7) | 13 (13)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Central nervous system infection (Infections and infestations) | 5 (6) | 5 (5)
Empyema (Infections and infestations) | 1 (1) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 106 (115) | 113 (125)
Sepsis (Infections and infestations) | 8 (8) | 9 (9)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 2 (2)
Tracheobronchitis (Infections and infestations) | 2 (2) | 4 (4)
Tracheostomy infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (6) | 3 (3)
Wound infection (Infections and infestations) | 5 (5) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 5 (5) | 8 (8)
Extradural hematoma (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (5)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural complication (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Shunt malfunction (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Subdural hemorrhage (Injury, poisoning and procedural complications) | 6 (7) | 4 (4)
Urethral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Bacterial test positive (Investigations) | 4 (4) | 4 (5)
Blood bilirubin increased (Investigations) | 4 (4) | 3 (3)
Cardiac enzymes increased (Investigations) | 2 (2) | 2 (2)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Cerebral salt-wasting syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 7 (7)
Hypovolemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cerebral hygroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 2 (2)
Brain edema (Nervous system disorders) | 22 (22) | 16 (17)
Brain injury (Nervous system disorders) | 10 (10) | 8 (8)
Cerebral hemorrhage (Nervous system disorders) | 8 (8) | 4 (4)
Cerebral venous thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrospinal fluid rhinorrhea (Nervous system disorders) | 1 (1) | 1 (1)
Chorea (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 6 (6) | 8 (9)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhage intracranial (Nervous system disorders) | 6 (6) | 12 (12)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 12 (12) | 8 (8)
Intracranial hypotension (Nervous system disorders) | 1 (1) | 0 (0)
Ischemic stroke (Nervous system disorders) | 5 (5) | 13 (13)
Neurological decompensation (Nervous system disorders) | 7 (7) | 11 (11)
Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 3 (3) | 0 (0)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1) | 3 (3)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 3 (3) | 3 (4)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 2 (2)
Impulsive behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 8 (9) | 7 (7)
Personality change (Psychiatric disorders) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 9 (9) | 7 (7)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 8 (8)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 6 (6)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 11 (11)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 11 (11)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 22 (22) | 16 (16)
Stridor (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Respite care (Social circumstances) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 2 (2) | 2 (2)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 2 (2) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 33 (36) | 27 (27)
Hemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 12 (12) | 5 (5)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone (N=442) | Placebo (N=440)
Anemia (Blood and lymphatic system disorders) | 8 (9) | 11 (12)
Coagulopathy (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 12 (13) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 7 (7)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 4 (4)
Bradycardia (Cardiac disorders) | 5 (6) | 10 (11)
Extrasystoles (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 4 (4) | 2 (2)
Tachycardia (Cardiac disorders) | 13 (13) | 8 (11)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 3 (3) | 2 (2)
Conjunctival oedema (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Mydriasis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (7) | 3 (3)
Adverse drug reaction (General disorders) | 1 (1) | 1 (1)
Catheter site hemorrhage (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1)
Edema peripheral (General disorders) | 1 (1) | 0 (0)
Infusion site edema (General disorders) | 12 (14) | 4 (5)
Infusion site erythema (General disorders) | 7 (7) | 3 (3)
Infusion site extravasation (General disorders) | 15 (16) | 9 (10)
Infusion site pain (General disorders) | 1 (1) | 1 (1)
Local swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 4 (4) | 2 (2)
Central nervous system infection (Infections and infestations) | 1 (1) | 2 (2)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 53 (54) | 49 (50)
Respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 14 (14) | 15 (15)
Vaginal infection (Infections and infestations) | 3 (3) | 2 (2)
Wound infection (Infections and infestations) | 1 (1) | 2 (2)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Heart injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Subdural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acid base balance abnormal (Investigations) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 0 (0)
Amylase increased (Investigations) | 2 (2) | 0 (0)
Bacterial test positive (Investigations) | 6 (6) | 2 (2)
Blood albumin decreased (Investigations) | 1 (1) | 2 (3)
Blood bicarbonate abnormal (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 12 (12) | 8 (8)
Blood calcium abnormal (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 2 (2)
Blood fibrinogen increased (Investigations) | 1 (1) | 0 (0)
Blood folate decreased (Investigations) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 7 (8) | 1 (1)
Blood magnesium abnormal (Investigations) | 0 (0) | 3 (3)
Blood osmolarity increased (Investigations) | 4 (4) | 3 (3)
Blood phosphorus abnormal (Investigations) | 0 (0) | 1 (1)
Blood potassium abnormal (Investigations) | 2 (2) | 4 (4)
Blood sodium abnormal (Investigations) | 2 (2) | 2 (2)
Blood urea increased (Investigations) | 2 (2) | 0 (0)
Cardiac enzymes increased (Investigations) | 1 (1) | 2 (2)
Drug level below therapeutic (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 2 (2) | 0 (0)
Full blood count abnormal (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 8 (8) | 8 (8)
International normalised ratio increased (Investigations) | 4 (4) | 1 (1)
Myoglobin blood increased (Investigations) | 1 (1) | 1 (1)
Prealbumin decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count abnormal (Investigations) | 2 (2) | 4 (4)
Acidosis (Metabolism and nutrition disorders) | 7 (7) | 11 (11)
Alkalosis (Metabolism and nutrition disorders) | 9 (9) | 8 (8)
Fluid overload (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hyperchloremia (Metabolism and nutrition disorders) | 7 (9) | 9 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (8) | 3 (3)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 5 (6) | 5 (5)
Hypernatremia (Metabolism and nutrition disorders) | 21 (21) | 29 (29)
Hyperphosphatemia (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 78 (83) | 101 (110)
Hypochloremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 72 (83) | 111 (129)
Hypomagnesemia (Metabolism and nutrition disorders) | 90 (101) | 94 (100)
Hyponatremia (Metabolism and nutrition disorders) | 29 (30) | 20 (21)
Hypophosphatemia (Metabolism and nutrition disorders) | 134 (145) | 134 (146)
Hypovolemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Propofol infusion syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 2 (2) | 4 (4)
Brain edema (Nervous system disorders) | 0 (0) | 3 (3)
Cerebral hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral venous thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrospinal fluid rhinorrhea (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 5 (5) | 9 (9)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
Hemorrhage intracranial (Nervous system disorders) | 3 (3) | 4 (4)
Ischemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Neurological decompensation (Nervous system disorders) | 1 (1) | 0 (0)
Paresis (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
VIth nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 1 (1) | 2 (2)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Impulsive behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 10 (11) | 10 (10)
Withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 7 (7)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 22 (24)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Artery dissection (Vascular disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 20 (22) | 13 (13)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)
Peripheral ischemia (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 74 (89) | 24 (27)
Thrombosis (Vascular disorders) | 2 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
The trial was stopped early for futility with respect to the primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No